CLINICAL TRIAL: NCT00757835
Title: 24-hour IOP Control With the Travoprost/Timolol Fixed Combination Compared With the Latanoprost/Timolol Fixed Combination, When Both Are Dosed in the Evening in Patients With Exfoliative Glaucoma
Brief Title: 24-hr IOP With Travoprost/Timolol Compared With Latanoprost/Timolol in XFG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A6219
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Glaucoma
Keywords: 24-hour IOP; exfoliative glaucoma; travoprost/timolol; latanoprost/timolol; fixed combinations
MeSH Terms: conditions — Glaucoma | interventions — Therapeutics; Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost/timolol therapy (Active Comparator): treatment with travoprost/timolol fixed combination drops once in the evening for 3 months. 24-hour pressure monitoring.
  Interventions: Drug: treatment with latanoprost/timolol fixed combination; Drug: latanoprost/timolol fixed combination drops
- Latanoprost/timolol therapy (Active Comparator): Treatment with latanoprost/timolol fixed combination for 3 months. 24-hour pressure monitoring.
  Interventions: Drug: treatment with latanoprost/timolol fixed combination; Drug: latanoprost/timolol fixed combination drops

INTERVENTIONS:
Drug: treatment with latanoprost/timolol fixed combination — dosing in the evening with the two fixed combinations
Drug: latanoprost/timolol fixed combination drops — once in the evening

SUMMARY:
A crossover, randomized, single-masked study which compares the short-term (3 months) 24-hour IOP control and safety of travoprost/timolol fixed combination given once in the evening, versus that of latanoprost/timolol fixed combination given once in the evening in patients with exfoliative glaucoma. The primary objective of this trial is to compare the quality of 24-hour IOP control after 3 months of chronic therapy with these two medications.

ELIGIBILITY:
Inclusion Criteria:

* Patient has XFG and is older than 29 years
* The IOP without treatment is greater than 25 mm Hg and lower than 40 mm Hg at baseline (2 readings at 10:00)
* Patient can be safely washed out without risk for significant deterioration
* Distance best corrected Snelen visual acuity better than 0.1
* No contraindication to prostaglandins or β-blockers
* No history of lack of response (<10% reduction) to any medication
* Patient can understand the instructions and comply to medications
* Open normal appearing angles
* No sign of ocular infection, except blepharitis, corneal abnormality that may affect IOP measurements etc

Exclusion Criteria:

* History of trauma, inflammation, surgery, past use of steroids (within 2 months), severe dry eyes and use of contact lenses
* Patient is a female of childbearing potential or lactating mother

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Travoprost/timolol fixed combination will demonstrate better quality of 24-hour IOP control than latanoprost/timolol | 3 months

SECONDARY OUTCOMES:
Incidence of side effects with the two medications | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios G Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, 1st University Department of Ophthalmology